CLINICAL TRIAL: NCT05949008
Title: Effect of Metformin ER With Hypocaloric Diet on Weight Loss in Overweight/Obese Patients With Increased Waist Circumference
Brief Title: Effect of Metformin, a Drug Used to Treat Diabetes, vs Placebo
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Vijaya Surampudi MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-001670
Record Dates: First submitted 2023-06-13; First posted 2023-07-17 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: NIDDM; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, controlled trial. All eligible participants will be randomly assigned to placebo or Metformin.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin Extended Release (ER) Oral Tablets (Experimental): This is a 24-week, randomized, double-blinded, two arm parallel clinical trial comparing metformin ER vs. placebo in combination with a hypocaloric diet (-500 kcal/day). 150 individuals with obesity and increased waist circumference will be randomized to taking metformin ER with hypocaloric diet or placebo with hypocaloric diet. All patients will receive dietary and exercise counseling with the intent of reducing their average caloric intake by 500 kcal/day.
  Interventions: Drug: Metformin Extended Release (ER) Oral Tablet
- Placebo (Placebo Comparator): Patients in the placebo arm will be randomized to placebo with hypocaloric diet. All patients will receive dietary and exercise counseling with the intent of reducing their average caloric intake by 500 kcal/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin Extended Release (ER) Oral Tablet — Metformin ER will be provided as 1000 mg capsules by Qingdao Baheal Pharmaceutical Co., Ltd. In addition to the active ingredient metformin HCl,each tablet contains the following inactive ingredients: Povidone, Sodium Lauryl Sulfate, Magnesium Stearate, Cellulose Acetate, Polyethylene Glycol (PEG 400, PEG 8000), Triacetin, Hypromellose, Titanium Dioxide, Polysorbate 80, Ferrosoferric Oxide, Shellac.
  Arms: Metformin Extended Release (ER) Oral Tablets
Drug: Placebo — Matching placebo will be provided as 1000 mg capsules
  Arms: Placebo

SUMMARY:
Metformin is a drug used to treat patients with diabetes. The aim of this study is to examine the effect of Metformin along with a low-calorie diet on obese and/or overweight adults with an increased waist measurement. In addition, the study also aims to look at the effect of the drug vs. placebo on quality of life and physical activity.

DETAILED DESCRIPTION:
Obesity is a growing epidemic in the United States. Weight gain is associated with an increased risk of developing life-threatening conditions such as high blood pressure or diabetes. Therefore, there is great interest in developing non-invasive treatments to help combat obesity. Currently, there are only few weight-loss drugs available for the treatment of obesity. In the more recent past, GLP-1 analogues (a type of non-insulin medication used to treat patients with diabetes) are being promoted as a new strategy to lose weight without major side effects however, with high costs and challenging supply chain issues.

This is a double-blinded, randomized study. This means that participants will be assigned to one of two groups. Participants will have a 1:1 chance of being assigned to receive either the study drug or a placebo (a capsule that does not contain the active ingredients). This assignment will be determined by chance. The process is similar to drawing cards or picking straws. This means your assignment to one of the groups is based on chance and not a medical decision made by the study doctor. In addition, neither participants nor the investigators will know what groups participants have been assigned to.

During this study, your participation will last up to 26 weeks (including screen) with a total of 8 clinic visits. Participants will undergo a total of 5 blood draws, blood samples will be taken at screen baseline and weeks 8, 16 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years at the time of signing informed consent.
* Body Mass Index (BMI) ≥ 27 kg/m2
* Waist circumference >40" for men, and >35" for women

Exclusion Criteria:

* A self-reported change in body weight > 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Diagnosed with T2D (HbA1c >7.5 (53 mmol/mol)
* Current use of insulin or oral medication of metformin, SU, SGLT2i, glitazone, DPP4 or GLP-1 agonist injections as single agent therapy or combination oral agents.
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of < 45 mL/min/1.73 m2 (< 60 ml/min/1.73 m2 in subjects treated with SGLT2i) according to CKDEPI creatinine equation as defined by KDIGO 201242 by the central laboratory at screening
* History of thyroid disease, but not taking medication or medication dosage changed one or more times over last 6 months (History of thyroid disease and on a stable dose of prescription medication for 6 months or longer is acceptable).
* History or lactic acidosis
* Liver problems
* Congestive heart failure
* History of alcoholism
* Recent surgery
* Heart attack, severe infection or stroke
* Any unstable medical conditions or terminal diagnosis
* Pregnancy or lactation
* Allergy and intolerance to metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve body weight reduction ≥5% from baseline | 24 Weeks
  Percent change in body weight reduction ≥5% from baseline (week 0) to week 24.
Change in total body weight from baseline | 24 Weeks
  Percent change in total body weight (TBW) from baseline (week 0) to week 24 in body weight.

SECONDARY OUTCOMES:
Change in total Body Mass Index (BMI) from baseline | 24 Weeks
  Change from baseline (week 0) to week 24 in: BMI
Percent change in body composition from baseline | 24 weeks
  Change from baseline (week 0) to week 24 - Body composition will be measured using a bioelectrical impedance analysis (BIA) scale. Measurements will include fat mass (kg), lean mass (kg), and body fat percentage. Data will be summarized as mean change from baseline to study endpoint for each group.
Change in waist circumference from baseline | 24 weeks
  Change from baseline (week 0) to week 24 in:Waist circumference (cm)
Change in insulin sensitivity from baseline | 24 Weeks
  Insulin sensitivity will be assessed using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), calculated from fasting glucose and fasting insulin levels. QUICKI (Quantitative Insulin Sensitivity Check Index) will be calculated using fasting glucose and insulin. The outcome will be reported as the change in QUICKI from baseline to Week 24.
Change in fasting blood lipids from baseline | 24 Weeks
  Change from baseline (week 0) to week 24 in Fasting blood lipids
Change in vascular function parameters (blood pressure and pulse wave velocity) | 24 weeks
  Vascular function will be assessed through two parameters:
  Systolic and diastolic blood pressure (mmHg)
  Pulse wave velocity (m/s) Each variable will be reported as a change from baseline to Week 24.
Change in inflammatory markers from baseline | 24 weeks
Change in daily dietary intake (calories and macronutrients) | 24 weeks
  Daily energy and macronutrient intake will be assessed using 3-day food records. The outcome includes:
  Total energy intake (kcal/day) Carbohydrate intake (g/day) Protein intake (g/day) Fat intake (g/day) Each variable will be reported as a change from baseline to Week 24.
Change in physical activity levels from baseline | 24 weeks
  Physical activity will be tracked using MyFitnessPal, which syncs data from wearable devices and user-logged exercise sessions. The following variables will be assessed:
  Average daily step count (steps/day) Weekly exercise duration (minutes/week), including structured physical activity Exercise frequency (days/week)
Change in quality of life from baseline | 24 weeks
  ● SF-36 QOL questionnaire
Change in glycemic control | 24 weeks
  Glycemic control will be assessed by measuring fasting glucose (mg/dL), fasting insulin (µIU/mL), and glycated hemoglobin A1c (reported as % and mmol/mol). All three measures will be obtained at baseline and Week 24. Each parameter will be reported as a change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Vijiya Surampudi, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No